CLINICAL TRIAL: NCT03537469
Title: Modulation of Long-Term Potentiation-Like Cortical Plasticity in the Healthy Brain With Low Frequency-Pulsed Electromagnetic Fields
Brief Title: Neuromodulation With Low Frequency-Pulsed Electromagnetic Fields
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, MAURO MAGONI, Head of U.O. Neurologia Vascolare, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NP-2322
Record Dates: First submitted 2018-04-29; First posted 2018-05-25 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Electromagnetic Fields; Neuronal Plasticity; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects and operators who performed TMS were blinded to the type of stimulation applied, we then employed a randomized double-blind sham-controlled crossover design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTU Mega 20 real device (Experimental): A single-session of real CTU Mega 20 on the corresponding primary right-hand motor area, using the real (magnetic field = 2 Tesla; intensity = 90 J; frequency of impulses = 7Hz; duration = 15 minutes) CTU Mega 20 device. This real stimulation provided a Low Frequency-Pulsed Electromagnetic Fields (LF-PEMFs).
  Interventions: Device: CTU Mega 20 real device
- CTU Mega 20 sham device (Sham Comparator): A single-session of sham CTU Mega 20 on the corresponding primary right-hand motor area (magnetic field = 0 Tesla; intensity = 0 J; frequency of impulses = 7Hz; duration = 15 minutes). The sham stimulation did not provide a Low Frequency-Pulsed Electromagnetic Fields (LF-PEMFs).
  Interventions: Device: CTU Mega 20 sham device

INTERVENTIONS:
Device: CTU Mega 20 real device — The CTU Mega 20 diamagnetic acceleration system discharges high-field magnetic impulses (with a duration of 5 ms and a period of 1000 ms), generating a magnetic field up to 2 Tesla, with a frequency of 7500 Hz in a volume of approximately 27 cm3.
  Arms: CTU Mega 20 real device
Device: CTU Mega 20 sham device — A CTU Mega 20 sham device (with an identical appearance to that of the real device) to avoid treatment identification by the patient or experimenter was used. Of course, the application of this sham device did not provide any magnetic field.
  Arms: CTU Mega 20 sham device

SUMMARY:
Non-depolarizing magnetic fields, like Low Frequency-Pulsed Electromagnetic Fields (LF-PEMFs) have shown the ability to modulate living structures, principally by influencing synaptic activity and ion channels on cellular membranes. Recently, the CTU Mega 20 device was presented as a molecular accelerator, using energy up to 200 Joules and providing high-power (2 Tesla) pulsating fields with a water-repulsive (diamagnetic) action and tissue biostimulation. The investigators tested the hypothesis that LF-PEMFs could modulate long-term corticospinal excitability in healthy brains by applying CTU Mega 20®. Ten healthy subjects without known neurological and/or psychiatric diseases entered the study. A randomized double-blind sham-controlled crossover design was employed, recording TMS parameters (amplitude variation of the motor evoked potential as index of cortical excitability perturbations of the motor system) before (pre) and after (post +0, +15, +30 min) a single CTU Mega 20 session on the corresponding primary right-hand motor area, using a real (magnetic field = 2 Tesla; intensity = 90 J; impulse frequency = 7Hz; duration = 15 minutes) or sham device. A two-way repeated measures ANOVA with TIME (pre, post +0, +15, +30 min) and TREATMENT (real vs sham stimulation) as within-subjects factor was applied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18 and 35 years

Exclusion Criteria:

* Known neurological or psychiatric diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Cortical Excitability change across time | Baseline and after 15, and 30 minutes
  Motor evoked potential (MEP) amplitude registered by TMS after sham or real stimulation at different time points, evaluating the differences among timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Magoni, MD, Principal Investigator — U.O. Neurologia Vascolare, Azienda Ospedaliera Spedali Civili, Brescia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Premi E, Benussi A, La Gatta A, Visconti S, Costa A, Gilberti N, Cantoni V, Padovani A, Borroni B, Magoni M. Modulation of long-term potentiation-like cortical plasticity in the healthy brain with low frequency-pulsed electromagnetic fields. BMC Neurosci. 2018 Jun 13;19(1):34. doi: 10.1186/s12868-018-0434-z. PMID 29895259